CLINICAL TRIAL: NCT05872217
Title: VIRTUAL REALITY TECHNOLOGY FOR UPPER EXTREMITY REHABILITATION OF CHILDREN WITH UNILATERAL CEREBRAL PALSY
Brief Title: VIRTUAL REALITY TECHNOLOGY FOR CEREBRAL PALSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VRapeutic software
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cerebral Palsy
Keywords: virtual reality; cerebralpalsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: intervention Control Group: Children in this group will receive conventional UE therapeutic program for about 60 minutes/3session per week.
  Children in this group will receive the same conventional UE therapeutic program as control group in addition to virtual reality session using fully-immersive VRapeutic software gaming technology (Archeeko module) for 30 min/3sessions/week for 8 weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A prospective randomized controlled trial of pre-post study design with two months follow-up evaluation will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): • This group will receive conventional UE therapeutic program for 60 minutes each session including:
  * Exercises based on neurodevelopment technique .
  * Gentle manual stretching
  * Weight-bearing exercises for 10minutes for UE from prone lying, side sitting and quadriped position .
  * Strengthening exercises for 10 minutes for muscles of UE as push-up from prone lying position, quadriped position, 3 point exercise, walk on hand, climbing, hanging on a bar, squeeze stress balls, cutting usescissors to strengthen hand .
  * Goal directed training for 10 minutes the child will practice specific tasks that are needed for everyday life and which they find a challenge like (3 daily tasks as cleaning mirror, dressing and undressing, using pen and ruler to draw shapes, brushing teeth .
  * Fine motor activities as reach, grasp, carry and release activities.
  Interventions: Other: conventional upper extremity therapeutic program
- study group (Experimental): Children in this group will receive the same conventional UE therapeutic program as control group for 60 minutes in addition to virtual reality session using VRapeutic software gaming technology, Archeeko module (figure 3) for 30 min/3 sessions/week for 8 weeks
  Interventions: Other: conventional upper extremity therapeutic program; Other: full immersive VRapeutic software gaming technology

INTERVENTIONS:
Other: conventional upper extremity therapeutic program — • This group will receive conventional UE therapeutic program for 60 minutes each session including:
  * Exercises based on neurodevelopment technique .
  * Gentle manual stretching for tight muscles of the affected UE from proximal to distal segments for 5minutes.
  * Weight-bearing exercises for 10minutes for UE from prone lying, side sitting and quadriped position.
  * Strengthening exercises for 10 minutes for muscles of UE as push-up from prone lying position, quadriped position, 3 point exercise, walk on hand, climbing, hanging on a bar, squeeze stress balls, cutting usescissors to strengthen hand .
  * Goal directed training for 10 minutes the child will practice specific tasks that are needed for everyday life and which they find a challenge like (3 daily tasks as cleaning mirror, dressing and undressing, using pen and ruler to draw shapes, brushing teeth .
  * Fine motor activities as reach, grasp, carry and release activities.
Other: full immersive VRapeutic software gaming technology — • Children in this group will receive the same conventional UE therapeutic program as control group for 60 minutes in addition to virtual reality session using VRapeutic software gaming technology, Archeeko module (figure 3) for 30 min/3 sessions/week for 8 weeks
  Arms: study group

SUMMARY:
The VRapeutic (Full-immersive game-based therapy) is new therapeutic Egyptian software. It has the potential to provide intensive, repetitive, and task-oriented training. It may increase children's motivation, enjoyment, active social participation. Children with UCP may experience varieties of associated health conditions as difficulty of movement, instability of postural balance, difficulty of motor planning and control which impact on UE function.

DETAILED DESCRIPTION:
Ethical statement this study was approved by institutional Review Board of the faculty of physical therapy ,cairo university .Egypt (no.P.T.REC/012/004237) .

Study Design A prospective randomized controlled trial of pre-post study design with two months follow-up evaluation will be used.

Sample size estimation

will be conducted to determine the number of recruited children. G*POWER statistical software (version 3.1.9.2) will be used using α=0.05, power 80% allocation ratio N2/N1 =1.

Randomization The selected children will be assigned by simple randomization via closed envelopes into two equal groups (control and study); the envelope will be contained a letter indicating whether the child will be assigned to the control or to the study group.

ELIGIBILITY:
Inclusion Criteria:

* • Their ages will range from of 6 to 10 years.

  * Both genders will be included.
  * Their degree of spasticity will range from 1 to 1+ according to the Modified Ashworth Scale (Meseguer et al., 2018).
  * Their motor function will be at level I according to Gross Motor Function Classification System (Palisano et al., 2008).
  * They will be able to understand and follow the instructions.

Exclusion Criteria:

* Exclusion Criteria:

Children will be excluded from the study if they have any of the following criteria:

* Epilepsy.
* Visual or hearing problems.
* Musculoskeletal fixed deformity in upper limbs, lower limbs or spine.
* Orthopedic surgery on the involved UE.
* Botulinum toxin therapy for the affected UE within the past 6 months or within the study period.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
rang of motion | period of treatment will be 2 succssive months
  The IMU sensors will be used to detect changes in angular displacement of child arm, forearm (which allow 3D analysis of movements in three planes X.Y.Z), speed and direction.
  Placement of Sensors: Two sensors will be placed on the affected side, one around the arm distal to shoulder joint and the other around the forearm distal to elbow joint. The third sensor will be placed around the trunk.
  The child will be in standing position with head in neutral position, trunk erect. The examiner will ask the child to perform functional task in form of (reaching forward toward targets placed on wall in multilevel, hand over head).
• ABILHAND-Kids questionnaire | period of treatment will be 2 succssive months
  will be administrated on an interview basis, the child will be asked to estimate their perception of the level of difficulty that faces during the performance of each activity in the list on a three-point ordinal scale of impossible, difficult, easy. Activities will be presented in random order to avoid any systematic effect. Activities not attempted in the last 3 months are not scored and are entered as missing responses (tick the question mark).

CONTACTS AND LOCATIONS:
Overall Officials: Eman I Elhadidy, Study Chair — Cairo University; Maya G Abd elwahab, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No